CLINICAL TRIAL: NCT02385916
Title: A Randomised, Double Blind, Placebo Controlled, Cross-over Trial Evaluating the Effects of EstroSense®/MD (PNO) vs Placebo in Increasing 2:16α Ratio and Improving the Estrogen Profile in Females
Brief Title: The Effects of EstroSense®/MD vs Placebo in Improving the Estrogen Profile in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Tim Green, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: H15-00279
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2016-05

CONDITIONS: Estrogen Profile
Keywords: EstroSense; estrogen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EstroSense®/MD (Experimental): 3 capsules per day during the study period
  Interventions: Other: Placebo
- Placebo (Placebo Comparator): 3 capsules per day during the study period
  Interventions: Other: EstroSense®/MD

INTERVENTIONS:
Other: EstroSense®/MD — A natural product already approved by Health Canada
  Arms: Placebo
Other: Placebo — Placebo
  Arms: EstroSense®/MD

SUMMARY:
According to the Canadian Cancer Society, 1 in 9 Canadian women will develop breast cancer in her lifetime and 1 in 30 will die. The single greatest risk factor of breast cancer is poor estrogen metabolism. EstroSense®/MD is a natural health product that promotes and supports healthy estrogen metabolism. It may increase the ratio of "good estrogen" to "bad estrogen" and potentially reducing the risk of breast cancer. For this proposed study, the investigators will be examining the effect of EstroSense®/MD compared to placebo, on estrogen metabolism in 120 women.

DETAILED DESCRIPTION:
This randomised, double blind, placebo controlled, crossover trial will evaluate the effects of daily consumption of EstroSense®/MD on estrogen profile in female subjects. 120 consenting women will be enrolled (randomised) to participate in this study. Potential subjects will be recruited by advertisements placed on notice boards around the university and at local naturopath clinics. Advertisements may also be placed in local newspapers. The study consists of four clinic visits. Individuals who are interested in participating will be asked to contact the study coordinator to schedule their first clinic visit (Visit 1). At Visit 1 the participant will be given information about the study and be given an opportunity to ask about the study. Those women who are still interested in participating will be asked to sign a consent form. Once consent if obtained screening and baseline data collection will begin. If eligible, participants will be scheduled to return to the clinic 19-21 days after the beginning of their last or next menstruation for Visit 2. At Visit 2 baseline data collection will continue followed by random assignment to an intervention sequence. All participants will be given and instructed to consume 3 capsules per day of EstroSense®/MD or Placebo for three menstrual cycles. After consuming the study intervention for 3 cycles, the participant will be asked to return to the clinic (19-21 days after the start of their third menstruation) for Visit 3. At Visit 3 data will be collected and participants will be crossed over to the other treatment for three more cycles. After 3 menstrual cycles (19-21 days after the start of their third menstruation) the participant will return to the clinic for Visit 4 for final data collection. Visit 4 marks the end of the study. Participants will also be provided with a diary throughout the study to record supplement use and any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* a woman
* 20-50 years of age
* willing to follow the treatment protocol, study visits and investigations as required by the study.

Exclusion Criteria:

* are on some certain medications that can interfere with the study such as hormone replacement medications (except birth control), anticoagulants, antiplatelet medications, digoxin, diuretics and breast cancer medications,
* are taking any natural health products that can alter estrogen levels, such as indole-3-carbinol, flaxseed, borage and primrose oil,
* smoke,
* are pregnant or nursing,
* have cancer,
* fibrocystic breast disease,
* family history of ovarian cancer,
* low estrogen or symptoms of low estrogen,
* stomach ulcers or excess stomach acids,
* a known iron deficiency,
* gall stones or bile duct obstruction,
* stomach ulcers or excess stomach acids,
* and or have a history of or known liver disease, kidney disease, thyroid disorders, or adrenal diseases.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Changes in urinary 2:16α Ratio | At baseline, 3 months, 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Green T, See J, Schauch M, Reil J, Glover M, Brix J, Gerry A, Li K, Newman M, Gahler RJ, Wood S. A randomized, double-blind, placebo-controlled, cross-over trial to evaluate the effect of EstroSense(R) on 2-hydroxyestrone:16alpha-hydroxyestrone ratio in premenopausal women. J Complement Integr Med. 2022 Oct 6;20(1):199-206. doi: 10.1515/jcim-2022-0301. eCollection 2023 Mar 1. PMID 36201753